CLINICAL TRIAL: NCT01517490
Title: Retinal Adaptation to Intensified Insulin Therapy and Bariatric Surgery in Patients With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Oliver Niels Klefter, Principal Investigator, Glostrup University Hospital, Copenhagen
Other Study IDs: Klefter1
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Insulin Infusion Systems; Bariatric Surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Type 1 Insulin Pump: Patients with type 1 diabetes starting insulin pump treatment
  Interventions: Other: Insulin pump
- Type 1 conventional therapy: Patients with type 1 diabetes continuing treatment with multiple daily insulin injections.
  Interventions: Other: Multiple daily insulin injections
- Type 2 Bariatric surgery: Patients with type 2 diabetes who are enrolled in pre-operative weight loss protocol prior to bariatric surgery.
  Interventions: Procedure: Bariatric surgery
- Type 2 conventional: Severely obese patients with type 2 diabetes who are to continue with non-surgical treatments of diabetes and obesity and with no planned bariatric surgery.
  Interventions: Other: Medical therapy for type 2 diabetes
- Type 1 insulin pumpe follow-up: Patients with type 1 diabetes previously followed in an observational study with electrophysiological and psychophysical measures of retinal function.
  Interventions: Other: Insulin pump
- Healthy: Healthy volunteers.

INTERVENTIONS:
Other: Insulin pump — Insulin pump therapy
  Groups: Type 1 Insulin Pump; Type 1 insulin pumpe follow-up
Other: Multiple daily insulin injections — Multiple daily insulin injections
  Groups: Type 1 conventional therapy
Procedure: Bariatric surgery — Pre-operative weight loss and bariatric surgery.
  Groups: Type 2 Bariatric surgery
Other: Medical therapy for type 2 diabetes — Medical glucose-lowering therapy and non-surgical weight-lowering interventions.
  Groups: Type 2 conventional

SUMMARY:
Retinal function is highly dependent on the glucose supply. Thus, functional adaptations occur in response to both acute and long-term changes in glycaemia.

The purpose of this study is to examine functional and metabolic aspects of retinal adaptation to long-lasting changes in glycaemic control in patients with diabetes. The adaptational phenomena will be characterized by electroretinography, dark adaptation, measures of retinal perfusion and oximetry as well as diabetic retinopathy grading and (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes and suboptimal metabolic regulation.
* Patients with type 2 diabetes and suboptimal metabolic regulation.

Exclusion Criteria:

* Significant cataract
* Glaucoma
* Proliferative diabetic retinopathy fulfilling ETDRS treatment criteria.
* Clinically significant macular edema fulfilling ETDRS treatment criteria.
* Age-related macular degeneration
* Prior surgery to the eye
* Other serious eye disease
* Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with type 1 diabetes and suboptimal metabolic regulation which is to be optimized by insulin pump therapy.
  30 patients with type 1 diabetes and suboptimal metabolic regulation in whom insulin pump therapy is not planned.
  20 patients with type 2 diabetes and suboptimal metabolic regulation who are enrolled in a pre-operative weight lowering protocol prior to bariatric surgery.
  20 patients with type 2 diabetes and suboptimal metabolic regulation who are not enrolled in treatment protocols relating to bariatric surgery.
  17 patients with type 1 diabetes on insulin pump therapy who were previously followed in an observational study of retinal function.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in dark adaptation kinetics and threshold values, amplitudes/implicit times, retinal vessel diameters, perfusion velocity and oximetry. | Baseline, 1 week, 1 month, 4 months, 7 months, 12 months, 18 months, 24 months, 42 months
Changes in visual acuity, diabetic retinopathy grading and OCT | Baseline, 1 week, 1 month, 4 months, 7 months, 12 months, 18 months, 24 months, 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klefter, MD, Principal Investigator — Glostrup UH; Michael Larsen, Professor, DMSci, Study Director — Glostrup UH
Locations (1):
- Department of Ophthalmology, Glostrup Hospital, Glostrup Municipality, Denmark